CLINICAL TRIAL: NCT06906809
Title: A Phase 1, Open-label, Fixed-sequence, Crossover Study to Investigate the Effect of Coadministration of the CYP3A Inducer Phenytoin and the CYP3A Inhibitor Itraconazole on the Pharmacokinetics of BGB-16673 in Healthy Participants
Brief Title: Effect of Phenytoin or Itraconazole on How BGB-16673 is Absorbed and Removed From the Body in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BGB-16673-105
Record Dates: First submitted 2025-03-26; First posted 2025-04-02 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-10

CONDITIONS: Healthy Volunteers
Keywords: BGB-16673; Drug-drug interactions; Pharmacokinetics
MeSH Terms: interventions — Itraconazole; Phenytoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part A: BGB-16673 + Phenytoin (CYP3A Inducer) (Experimental): Participants will receive multiple doses of Phenytoin to determine its effect on BGB-16673
  Interventions: Drug: BGB-16673; Drug: Phenytoin
- Part B: BGB-16673 + Itraconazole (CYP3A Inhibitor) (Experimental): Participants will receive multiple doses of Itraconazole to determine its effect on BGB-16673
  Interventions: Drug: BGB-16673; Drug: Itraconazole

INTERVENTIONS:
Drug: BGB-16673 — Administered orally
Drug: Itraconazole — Administered orally
  Arms: Part B: BGB-16673 + Itraconazole (CYP3A Inhibitor)
Drug: Phenytoin — Administered orally
  Arms: Part A: BGB-16673 + Phenytoin (CYP3A Inducer)

SUMMARY:
The purpose of this study is to investigate the effect of coadministration of phenytoin or itraconazole on the pharmacokinetics of BGB-16673 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, of any race, between 18 and 65 years of age
* In good health, as determined by no clinically significant findings from medical history,12- lead ECG and vital signs measurements, physical examination and clinical laboratory evaluations
* Body mass index between 18.0 and 32.0kg/m2, inclusive

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator or designee.
* Evidence of any infections (bacterial, viral, fungal, parasitic) within 4 weeks prior to the first dose of study drug, as determined by the investigator (or designee).
* History of malignancy, except for appropriately treated carcinoma in situ of the cervix or nonmelanoma skin carcinoma not requiring ongoing systemic treatment.
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair are allowed).
* Participants who have acute gastrointestinal symptoms at the time of screening and or/admission (eg, nausea, vomiting, diarrhea, or heartburn).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2025-04-03 (Actual); Primary Completion 2025-10-13 (Actual); Study Completion 2025-10-13 (Actual)

PRIMARY OUTCOMES:
Part A and Part B: Area Under the Concentration-time Curve from Time 0 Extrapolated to Infinity (AUC0-∞) of BGB-16673 | Part A: Day 1 and Day 20; Part B: Day 1 and Day 17
Part A and Part B: Area Under the Concentration-time Curve from Time 0 to the Time of the Last Quantifiable Concentration (AUC0-tlast) of BGB-16673 | Part A: Day 1 and Day 20; Part B: Day 1 and Day 17
Part A and Part B: Maximum Observed Concentration (Cmax) of BGB-16673 | Part A: Day 1 and Day 20; Part B: Day 1 and Day 17

SECONDARY OUTCOMES:
Part A and Part B: Time of the Maximum Observed Concentration (Tmax) of BGB-16673 | Part A: Day 1 and Day 20; Part B: Day 1 and Day 17
Part A and Part B: Apparent Terminal Elimination Half-life (t1/2) of BGB-16673 | Part A: Day 1 and Day 20; Part B: Day 1 and Day 17
Part A and Part B: Apparent Total Clearance (CL/F) of BGB-16673 | Part A: Day 1 and Day 20; Part B: Day 1 and Day 17
Part A and Part B: Apparent Volume of Distribution During the Terminal Phase (Vz/F) of BGB-16673 | Part A: Day 1 and Day 20; Part B: Day 1 and Day 17
Part A and Part B: Number of Participants with Adverse Events (AEs) | Up to approximately 36 days
  Safety will be assessed by monitoring and recording of all treatment emergent adverse events (AEs) graded by National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0
Part A and Part B: Number of Participants with Clinically Significant Laboratory Values | Up to approximately 36 days
Part A and Part B: Number of Participants with Clinically Significant Electrocardiogram (ECG) results | Up to approximately 36 days
Part A and Part B: Number of Participants with Clinically Significant Vital Sign Measurements | Up to approximately 36 days

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (1):
- Fortrea Clinical Research Unit Inc, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/